CLINICAL TRIAL: NCT06102967
Title: Correlation Between Intraoperative Electroencephalographic Signatures and Postoperative Delirium in Preoperative Frail Elderly Patients Undergoing
Brief Title: EEG Characteristics and Postoperative Delirium
Status: Completed | Type: Observational
Sponsor: Zhuo Liu (Other Government)
Responsible Party: Sponsor-Investigator, Zhuo Liu, Principal Investigator, The First Hospital of Qinhuangdao
Organization: The First Hospital of Qinhuangdao (Other Government)
Other Study IDs: lzh123456
Record Dates: First submitted 2023-10-09; First posted 2023-10-26 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Delirium; Cognitive Function Abnormal; PSI; Frailty
MeSH Terms: conditions — Emergence Delirium; Cognition Disorders; Frailty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-delirious group: No postoperative delirium occurred
- Delirious group: Postoperative delirium occurs
  Interventions: Behavioral: delirium

INTERVENTIONS:
Behavioral: delirium — Evaluation of delirium using the ICU Patient Ambiguity Assessment Form (CAM-ICU) 1 day, 2 days, 3 days, and 7 days after surgery
  Groups: Delirious group

SUMMARY:
The goal of this [type of study: observational study ] is to [compare Energy differences in various bands of intraoperative electroencephalogram in elderly patients with postoperative delirium and non delirium.] in [describe participant population selected 69 patients who underwent laparoscopic radical surgery for colorectal cancer on a selective basis]. The main question[s] it aims to answer are:

• [Is there any difference in the spectral range of EEG between POD patients and non POD patients] Participants will [Cognitive.•Postoperative delirium.•Preoperative weakness.]

DETAILED DESCRIPTION:
The goal of this [type of study: observational study ] is to [compare Correlation between EEG data and postoperative delirium in elderly patients undergoing colorectal cancer radical surgery under preoperative frailty monitoring.] in [describe participant population selected 69 patients who underwent laparoscopic radical surgery for colorectal cancer on a selective basis]. The main question[s] it aims to answer are:

• [Is there any difference in the spectral range of EEG between POD patients and non POD patients] Participants will [Sedline EEG monitoring electrodes were placed 1cm above the eyebrows on both sides of the patient and at the temples on both sides, and were continuously monitored from the start of anesthesia in the operating room until the end of the surgery.Pay close attention to the vital signs and wait for the patient to fully recover and the vital signs to basically return to the preoperative level before returning to the ward.•Assessment of cognitive function using the Mini Mental State Scale (MMSE) 1 day before surgery and 7 days after surgery.•Preoperative assessment of frailty using the frailty screening scale.•Assess delirium using the ICU Patient Ambiguity Assessment Form (CAM-ICU) 1 day, 2 days, 3 days, and 7 days after surgery.].

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* The preoperative Frailty Scale (FRAIL) assessed frailty
* The patient or his/her family is informed about the study and signs an informed consent form

Exclusion Criteria:

* Serious insufficiency of heart, liver, kidney and other functions
* Those with a history of psychiatric or neurological illness, long-term use of psychotropic drug
* History of cerebrovascular disease, brain trauma, or surgery
* The patient was allergic to coupler or unable to place electrodes on the head
* The patient was unable to complete the scale assessment as required.Patients with severe attention to hearing impairment were unable to complete the interview
* The patient was diagnosed with delirium before surgery

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing laparoscopic radical surgery for colorectal cancer on a scheduled basis.Age ≥ 65 years old, regardless of gender; ASA grading I to III; The preoperative frailty scale (FRAIL) was evaluated as frailty; The patient or their family members voluntarily sign an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium | 1 day, 2 days, 3 days, and 7 days after surgery
  Assessing delirium using the ICU Patient Ambiguity Assessment Form (CAM-ICU)
EEG power of each band | During the procedure
  Recording frontal lobe electroencephalogram using a sedline root monitor (Masimo, Crop)
The number of minutes of suppression assessed by visual analysis of the EEG | Throughout the operation
  The burst suppression time was calculated by EEG visual analysis

CONTACTS AND LOCATIONS:
Overall Officials: Qinshuang Liu, master, Study Director — The First hosptial of Qinhuangdao; Zhaoheng Li, master, Study Chair — The First hosptial of Qinhuangdao
Locations (1):
- The first hospital of Qinhuangdao, Qinhuangdao, Hebei, China

IPD SHARING:
Plan to Share IPD: No